CLINICAL TRIAL: NCT03763214
Title: Randomized Comparative Study of Novel PTFE-coated Stents (Hilzo) Versus Standard Silicone-coated Metal Stents (cSEMS) in Distal Malignant DHC Stenosis
Brief Title: PTFE Stents for Treatment of Malignant Biliary Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Vermehren (Other)
Collaborators: Robert Bosch Medical Center (Other); Klinikum Stadt Hanau (Other)
Responsible Party: Sponsor-Investigator, Johannes Vermehren, Record Keeper, Clinical Professor, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWGUHMED1-009
Record Dates: First submitted 2018-05-14; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Bile Duct Stricture; Bile Duct Cancer; Pancreas Cancer
Keywords: metal stent; biliary stricture; stenting
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms | interventions — Stents

STUDY DESIGN:
Intervention Model Description: Randomized, two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stenting with PTFE-coated stent (HILZO) (Experimental): The bile duct is stented with a PTFE-coated stent by duodenoscopy to allow bile duct flow
  Interventions: Device: Stenting with PTFE-coated stent (HILZO)
- Stenting standard silicone coated stent (Active Comparator): The bile duct is stented with a standard silicone-coated stent by duodenoscopy to allow bile duct flow
  Interventions: Device: Stenting with PTFE-coated stent (HILZO)

INTERVENTIONS:
Device: Stenting with PTFE-coated stent (HILZO) — Placing a metal stent in the biliary tract by duodenoscopy

SUMMARY:
In this randomized trial two two self-expanding metal stents (SEMS) for treatment of malignant biliary strictures are investigated.

A newly developed PTFE (Polytetrafluorethylen) (Teflon) stent is tested versus standard covered metal stents. PFTE (Teflon) coating promises improved formability over standard silicone-coated stents, easier removal through the soft surface, and significantly reduced tumor growth through the impermeable surface.

DETAILED DESCRIPTION:
ERCP (endoscopic retrograde cholangiopancreatography) is the standard method of treating diseases in the biliopancreatic system and the treatment goal is achieved in a very high proportion of the studies. The ERCP is based on the indirect imaging of the bile ducts by injection of contrast medium, which is visualized in X-ray fluoroscopy. Furthermore, the probing of the bile ducts by means of wire and direct interventions within the bile duct system is possible.

Malignant biliary strictures are caused by various, usually cholangiocellular or pancreatic tumors, whose surgical therapy is complex and often impossible due to advanced disease. Tumors of the papillae, lymphomas and lymph node metastases can also lead to stenosis of the extra hepatic bile ducts.

The outcome of patients with malignant biliary strictures is poor, most are already presenting with advanced disease because early symptoms are rare. In particular, the above-mentioned cholangiocellular carcinomas and pancreatic carcinomas are often resectable only in its early form with high recurrence rates. Furthermore, then only palliative concepts are possible. Various studies have shown that stenting of the biliary tract with drainage of more than 50% of the liver volume improves survival. Metal stents seem to be superior to plastic stents at a slightly higher cholangitis rate. It is therefore considered standard therapy to palliatively treat these patients with more than 3 months of life expectancy using a metal stent.

Two types of stents are currently in use, plastic stents and self-expanding metal stents (SEMS). These in turn are coated (cSEMS) and uncoated (uSEMS). In distal malignant stenosis, both cSEMS and uSEMS can be used, with a higher patency rate for cSEMS and a longer duration of uSEMS retention. The disadvantage of the uSEMS is the tumor ingrowth in the stents and the possibility of re-stenosis. Various studies have shown that metal stents are associated with better bile duct drainage and better retention time compared to plastic stents and have fewer early complications, however, a consensus regarding a survival advantage with metal stents has not yet been substantiated, with the data showing a positive trend. Since metal stents, unlike plastic stents, do not need to be changed, a significant advantage for the patient is the significant reduction in endoscopic examinations and associated hospitalization and complication rates.

PTFE stents are a new development that should significantly reduce tumor ingrowth into the stent and, in particular, allow for a significantly reduced stent migration rate. PFTE (Teflon) coating promises improved formability over standard silicone-coated stents, easier removal through the soft surface, and significantly reduced tumor growth through the impermeable surface. At both ends of the stents are "tulips" which are coated with silicone. This in turn reduces the rate of stent closure by sludge, and in particular, the otherwise very high rate of stent migration should be significantly reduced.

ELIGIBILITY:
Inclusion Criteria:

• Indication for the palliative metal-stent system for malignant stenosis of the distal DHC (bile duct tumors, pancreatic carcinoma, papillary carcinoma, lymphoma, lymph node metastases in the hilum)

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Contraindication to an endoscopic examination
* Life expectancy under 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Stent migration | 12 month
  Rate of stent migrations

SECONDARY OUTCOMES:
Stent dysfunction (re-stenosis) | 12 month
  Stenosis of stent with necessity to do duodenoscopy again
Number of ERCPs in one year | 12 month
  Count of the number of duodenoscopy the patients undergo
Survival rate | 12 month
  Survival of patientes 12 month after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany